CLINICAL TRIAL: NCT07233993
Title: A Randomised, Cross-over, Double-blind, Sham-Controlled Superiority Trial of UltraSound-Guided Versus Non-Ultrasound-Guided Botulinum TOxin Injections in Cervical DYstonia
Brief Title: UltraSound-Guided Versus Non-Ultrasound-Guided Botulinum Toxin Injections in Cervical Dystonia [CUSTODY]
Acronym: CUSTODY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CUSTODY
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Cervical Dystonia
Keywords: Cervical dystonia; Idiopathic cervical dystonia; Botulinum toxin; BoNT injections; Ultrasound-guided injections; Anatomical landmark; Quality of life; Motor symptoms; Non-motor symptoms
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, double-blind, sham-controlled, cross-over clinical trial. Participants with idiopathic cervical dystonia will receive both ultrasound-guided and non-ultrasound-guided botulinum toxin injections in two treatment periods, serving as their own control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to the injection technique. Injectors cannot be blinded for practical reasons. To maintain blinding, the ultrasound device will be present in all procedures. For participants randomized to the non-ultrasound group, the ultrasound probe will be positioned but the device screen will be turned off, so that the procedure appears identical to an ultrasound-guided injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided BoNT Injections (Experimental): Participants receive botulinum toxin type A injections into cervical muscles using real-time ultrasound guidance to visualise target muscles and surrounding structures
  Interventions: Procedure: Ultrasound-guided botulinum toxin injection; Procedure: Non-ultrasound-guided botulinum toxin injection
- Non-Ultrasound-Guided BoNT Injections (Sham Comparator): Participants receive botulinum toxin type A injections into cervical muscles using anatomical landmarks, without ultrasound guidance. The ultrasound device is present but the screen is turned off to maintain blinding.
  Interventions: Procedure: Ultrasound-guided botulinum toxin injection; Procedure: Non-ultrasound-guided botulinum toxin injection

INTERVENTIONS:
Procedure: Ultrasound-guided botulinum toxin injection — Botulinum toxin type A is injected into dystonic cervical muscles under real-time ultrasound guidance, allowing visualisation of target muscles and adjacent structures. Injections are performed according to standard clinical practice with a stable dose and scheme
Procedure: Non-ultrasound-guided botulinum toxin injection — Botulinum toxin type A is injected into dystonic cervical muscles using anatomical landmarks, without ultrasound guidance. To maintain blinding, the ultrasound device is present in all procedures, but the screen is turned off in this arm. Injections are performed according to standard clinical practice with a stable dose and scheme

SUMMARY:
Cervical dystonia is a condition that causes the neck muscles to tighten or spasm, leading to abnormal head positions and pain.

The main questions it aims to answer are:

* Do ultrasound-guided BoNT injections improve quality of life more than injections without ultrasound?
* Are ultrasound-guided injections as safe as injections without ultrasound?

Researchers will compare:

* BoNT injections with ultrasound guidance
* BoNT injections without ultrasound guidance (based only on body landmarks)

Participants will:

* Receive both types of injections during the study (one first, then the other)
* Complete questionnaires about quality of life, movement, pain, and mood
* Attend follow-up visits over about 8 months About 37 adults with cervical dystonia will take part. The study will take place at the Fondazione IRCCS Istituto Neurologico Carlo Besta in Milan, Italy.

DETAILED DESCRIPTION:
Cervical dystonia (CD) is the most common type of focal dystonia and is characterised by sustained or intermittent involuntary contractions of the neck muscles. These contractions lead to abnormal head postures and movements, frequently associated with pain and tremor, and have a major impact on quality of life.

The established treatment for CD is repeated intramuscular injections of botulinum toxin type A (BoNT-A), usually every 12 to 16 weeks. BoNT-A blocks acetylcholine release at the neuromuscular junction, producing a temporary and reversible chemodenervation of the target muscle. Clinical benefit generally appears within a few days, peaks after 2 to 4 weeks, and gradually wears off after 3 to 4 months, requiring repeated injections. Although this therapy is effective and safe, its clinical success largely depends on the accuracy of muscle targeting. Suboptimal precision in injections can lead to unsatisfactory outcomes, persistence of symptoms, or treatment discontinuation.

Several approaches are used in clinical practice to guide injections. The conventional method relies on palpation and anatomical landmarks, is widely available, and requires limited resources. However, it depends heavily on the injector's experience and may result in inaccurate targeting. Ultrasound (US) guidance, on the other hand, allows direct, real-time visualisation of the cervical muscles and adjacent structures. This technique may increase accuracy, optimise toxin distribution, and lower the risk of misplaced injections and adverse events.

Cadaveric studies have demonstrated higher accuracy of US-guided injections compared with landmark-based methods, and preliminary clinical studies suggest that US guidance may improve outcomes. However, these studies have been limited by small sample sizes, lack of randomisation, or non-blinded assessments. Robust evidence from randomised controlled trials is still lacking, and therefore the clinical superiority of US guided injectionsance remains uncertain.

US-guided injections also require additional equipment, time, and operator training. This may limit their widespread adoption in routine clinical practice unless a clear advantage over landmark-based injections is demonstrated. Addressing this knowledge gap is essential to inform clinical decisions and optimise the management of CD.

The present study has been designed to evaluate the impact of US-guided BoNT-A injections compared with injections based only on anatomical landmarks in adults with idiopathic CD. The primary objective is to determine whether US guidance provides superior improvements in quality of life. Secondary objectives include assessing the effects of the two techniques on motor and non-motor symptoms, as well as comparing their safety.

A total of approximately 37 participants with idiopathic cervical dystonia and a documented good response to prior BoNT-A therapy will be recruited at the Fondazione IRCCS Istituto Neurologico Carlo Besta in Milan, Italy. Each participant will undergo two treatment cycles, one with US guidance and one without, in randomised order. The duration of participation for each individual will be about 8 months. By directly comparing two widely used approaches, this trial will provide high-quality evidence to guide clinical practice and improve care for people with cervical dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years old
* Clinical diagnosis of Idiopathic Cervical Dystonia
* On a stable dose of other medications (if any) used for focal dystonia treatment (e.g. anticholinergics and benzodiazepines) for at least 3 months prior to screening and expected to be maintained throughout the study
* Treatment non-naïve to BoNT type A therapy for CD
* At least 4 months have passed between the last BoNT injection at screening
* Good clinical response to previous BoNT injections, on stable dosing and treatment scheme
* Informed Consent as documented by signature.
* Ability to perform study requirements (to attend assessment and treatments)

Exclusion Criteria:

* Diagnosis of other types of Cervical Dystonia (Inherited and Acquired)

  * Concomitant diagnosis of diseases that contraindicate the use of botulinum toxin, such as myasthenia gravis
  * Known hypersensitivity or allergy to Botulinum-A Toxin
  * Women who are pregnant or breast feeding
  * Intention to become pregnant during the study
  * Lack of safe contraception
  * Other clinically significant and unstable concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.).
  * Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
  * Participation in another study with investigational drug within the 30 days preceding and during the present study
  * Previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cervical Dystonia Impact Profile-58 (CDIP-58) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over desig
  Total score on the Cervical Dystonia Impact Profile (CDIP-58), a patient-reported outcome measure of quality of life in cervical dystonia. Score range: 0-100, with higher scores indicating greater impact on quality of life (worse outcome).

SECONDARY OUTCOMES:
Change in Toronto Western Spasmodic Torticollis Rating Scale - 2 (TWSTRS-2) | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  Total score on the Toronto Western Spasmodic Torticollis Rating Scale, 2nd edition (TWSTRS-2), a clinician-rated scale assessing severity, disability, and pain in cervical dystonia. Score range: 0-100, with higher scores indicating greater severity, disability, or pain (worse outcome).
Change in Psychiatric Screening Tool (TWSTRS-PSYCH) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  The TWSTRS-PSYCH assesses psychiatric comorbidity associated with cervical dystonia.
Change in Hospital Anxiety and Depression Scale (HADS) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  The HADS is a self-administered questionnaire that evaluates anxiety and depressive symptoms
Change in Pain Numerical Rating Scale (NRS) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  Difference in pain intensity measured with the NRS between baseline and 6 weeks after each injection, in both crossover
Change in Clinical Global Impression - Change (CGI-C) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  The CGI-C is a 7-point scale measuring overall clinical improvement.
Change in Patient Global Impression - Change (PGI-C) score | 6 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  Score on the Patient Global Impression of Change (PGI-C), a 7-point patient-reported scale reflecting the patient's impression of improvement. Score range: 1-7, with higher scores indicating greater improvement (better outcome).
Frequency of adverse events | From baseline to 16 weeks (±2 weeks) after each treatment, during both periods of the cross-over design.
  Number and type of any adverse events reported during both crossover periods. Safety will be assessed by comparing the frequency of adverse events between the two injection techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720